CLINICAL TRIAL: NCT06530524
Title: Pretherapy Botulinum Toxin to Reduce Radiation-related Xerostomia in Head and Neck Cancer
Brief Title: Pretreatment Botulinum Toxin in Head and Neck Cancer Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Lady Davis Institute (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Marco Mascarella, Principal Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROTOX
Record Dates: First submitted 2024-07-23; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Head Neck Cancer; Xerostomia Following Radiotherapy
Keywords: Head and Neck Cancer; Radiation induce xerostoma; botulinum toxin; salivary glands
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): The treating physician will perform the injection of normal saline under ultrasound guidance using a 30-gauge needle introduced into the salivary gland tissue. 30 units of normal saline will be infiltrated the major salivary glands at-risk.
  Interventions: Drug: Placebo
- onabotulinumtoxinA (Experimental): The treating physician will perform the injection of onabotulinumtoxinA under ultrasound guidance using a 30-gauge needle introduced into the salivary gland tissue. 30 units of onabotulinumtoxinA will be infiltrated the major salivary glands at-risk.
  Interventions: Drug: OnabotulinumtoxinA

INTERVENTIONS:
Drug: OnabotulinumtoxinA — Injection of onabotulinumtoxinA into the at-risk major salivary glands
  Arms: onabotulinumtoxinA
Drug: Placebo — Injection of normal saline into the at-risk major salivary glands
  Arms: Placebo

SUMMARY:
Head and neck cancer care, including tumors of the mouth, nose, throat and voice box, often requires radiation for cure to be achieved. Despite advances in radiation, 40% to 60% of patients experience a significant dry mouth (xerostomia) following radiotherapy. Several factors are associated with severe xerostomia including older age, advanced stage disease and tumor location. Currently, no pragmatic treatment strategy exists to reduce the risk of radiation-related xerostomia in patients with head and neck cancer. The investigators propose the use of a botulinum neurotoxin injected into the at-risk salivary glands before radiation as a strategy to preserve salivary gland function during radiation treatments and reduce xerostomia.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosis AJCC 8th edition Stage III/IVa mucosal head and neck squamous cell carcinoma requiring definitive radiotherapy (with or without chemotherapy).

Exclusion Criteria:

* Previous radiation to the head and neck
* Previous treatment for head and neck cancer
* Personal history of xerostomia
* Hypersensitivity to onabotulinumtoxinA
* Previous major salivary gland surgery
* Previous exposure to radioactive iodine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Xerostomia-related quality of life | Pretreatment, 6 and 12 months from treatment completion
  University of Washington Quality of Life questionnaire (higher score is better)

SECONDARY OUTCOMES:
Unstimulated salivary function using salivary gland scintigraphy | Pretreatment and 12 months from treatment completion
  Measurement of unstimulated salivary gland flow prior to initiation of therapy and at 12 months from completion of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No